CLINICAL TRIAL: NCT06232538
Title: A Prospective, Multi-centre, Single-blinded Study of UCAD for Diagnosing Benign or Malignant Gallbladder Diseases and Follow-up
Brief Title: UCAD for Diagnosing Benign or Malignant Gallbladder Diseases and Follow-up
Status: Active, not recruiting | Type: Observational
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Shanghai Zhongshan Hospital (Other); Ruijin Hospital (Other); Changhai Hospital (Other); Shanghai Changzheng Hospital (Other); Eastern Hepatobiliary Surgery Hospital (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); Jiangsu Provincial People's Hospital (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other); First Affiliated Hospital of Zhejiang University (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); Second Hospital of Jilin University (Other); West China Hospital (Other); Southwest Hospital, China (Other); Afﬁliated Hospital of North Sichuan Medical College (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: XH-24-001
Record Dates: First submitted 2024-01-22; First posted 2024-01-30 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Gallbladder Cancer
Keywords: diagnosis
MeSH Terms: conditions — Gallbladder Neoplasms; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA from bile in the gallbladder will be analyzed
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- gallbladder cancer
  Interventions: Diagnostic Test: The level of CNV
- benign gallbladder diseases
  Interventions: Diagnostic Test: The level of CNV

INTERVENTIONS:
Diagnostic Test: The level of CNV — The extracted DNA from bile will be analyzed by UCAD to determine the level of CNV. And the patient will be followed more than 1 year.

SUMMARY:
Copy number variation(CNV) refers to ongoing chromosome segregation errors throughout consecutive cell divisions. CNV is a hallmark of human cancer, and it is associated with poor prognosis, metastasis, and therapeutic resistance. Analyzing CNV of the DNA extracted from bile samples in gallbladder seems a promising method for diagnosing, monitoring, and predicting the prognosis of patients with gallbladder cancer. CNV can be assessed using experimental techniques such as bulk DNA sequencing, fluorescence in situ hybridization (FISH), or conventional karyotyping. However, these techniques are either time-consuming or non-specific. The investigators here intend to study whether a new method named Ultrasensitive Chromosomal Aneuploidy Detection (UCAD), which is based on low-coverage whole-genome sequencing, can be used to analyze CNV thus helping diagnose gallbladder cancer and assessing follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with gallbladder disease and planned to undergo surgery.
* Male or female patients aged >= 18 years.
* Participants signed informed consent form.

Exclusion Criteria:

* Participants had other tumor expect gallbladder cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with malignant biliary obstruction or participants in control group from February 2022 till the end of this study in 11 hospitals including Xinhua Hospital, Shanghai Zhongshan Hospital, Ruijin Hospital, Changhai Hospital, Shanghai Changzheng Hospital, Eastern Hepatobiliary Surgery Hospital, The First Affiliated Hospital of Xi'an Jiaotong University, Jiangsu Provincial Hospital, The Third Affiliated Hospital of Sun Yat-Sen University, Tianjin Medical University Second Hospital, First Affiliated Hospital of Zhejiang University
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
UCAD can be used as a diagnostic technology for gallbladder cancer with the sensitivity more than 90% | 2025
  Ultrasensitive chromosomal aneuploidy detection (UCAD) uses low-coverage whole-genome sequencing technology to detect DNA chromosomal instability in samples. By detecting DNA extracted from patients' bile and blood, bioinformatics can be used to analyze the differences in CNV between benign and malignant gallbladder diseases, and a prediction model for gallbladder cancer.

CONTACTS AND LOCATIONS:
Locations (1):
- Xinhua Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hieronymus H, Murali R, Tin A, Yadav K, Abida W, Moller H, Berney D, Scher H, Carver B, Scardino P, Schultz N, Taylor B, Vickers A, Cuzick J, Sawyers CL. Tumor copy number alteration burden is a pan-cancer prognostic factor associated with recurrence and death. Elife. 2018 Sep 4;7:e37294. doi: 10.7554/eLife.37294. PMID 30178746